CLINICAL TRIAL: NCT03292302
Title: A Phase 1a, Randomized, Double-blinded, Placebo-Controlled, Single Dose Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of ELX-02 in Healthy Adult Volunteers
Brief Title: Phase 1 Study of ELX-02 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eloxx Pharmaceuticals, Inc. (Industry)
Collaborators: SGS Life Sciences, a division of SGS Belgium NV (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EL-006
Record Dates: First submitted 2017-08-30; First posted 2017-09-25 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2019-10

CONDITIONS: Genetic Disease; Nonsense Mutation
Keywords: Translational read through
MeSH Terms: conditions — Genetic Diseases, Inborn | interventions — ELX-02

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Comparator Arm (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Active treatment (Active Comparator): ELX-02
  Interventions: Drug: ELX-02

INTERVENTIONS:
Drug: Placebo — Placebo comparator
  Arms: Placebo Comparator Arm
Drug: ELX-02 — Synthetic aminoglycoside
  Arms: Active treatment

SUMMARY:
Phase 1 Single Ascending Dose Study in Normal Healthy Volunteers

DETAILED DESCRIPTION:
This is a study in humans of ELX-02, an advanced synthetic aminoglycoside optimized as a translational read-through drug (TRID) for the treatment of genetic conditions caused by nonsense mutations. This is a classical Phase 1a study designed as a randomized, double-blinded, placebo-controlled, single dose escalation to evaluate the safety, tolerability and pharmacokinetics of ELX-02 in healthy adult volunteers.

ELIGIBILITY:
Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the study:

1. Be able and willing to provide written Informed Consent indicating that the subject has been informed of all pertinent aspects of the study.
2. Healthy female subjects and male subjects who, at the time of screening, are between the ages of 18 and 45 years, inclusive.

   Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure (BP) and pulse rate measurement, 12-lead electrocardiogram (ECG), and clinical laboratory tests.
3. Female subjects of nonchildbearing potential must meet at least one of the following criteria:

   * Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; post-menopausal status will be confirmed by a serum follicle-stimulating hormone level;
   * Have undergone a documented hysterectomy and/or bilateral oophorectomy;
   * Have medically confirmed ovarian failure. All other female subjects (including females with tubal ligations) will be considered to be of childbearing potential and may be enrolled if they have negative pregnancy tests at screening and admission day and agree to use a highly effective method of contraception for 14 days before study drug administration and 28 days after study drug administration. Female subjects of childbearing potential must agree to undergo repeated pregnancy tests. For highly effective methods of contraception include see Section 6.5.1.
4. Male subjects must be willing to use an effective method of contraception. They must agree to use a condom consistently and correctly, during the course of the study until 28 days after study drug administration.
5. Not using any prescription medication and dietary supplements within 30 days or 5 half-lives (whichever is longer) prior to the administration of study drug administration, except for contraceptives - nor be taking any over-the-counter (OTC) herbal or medicinal products. As an exception, acetaminophen/paracetamol may be used at doses of ≤ 2 g/day. Aspirin and non steroidal anti inflammatory drugs (NSAIDs) should not be administered within 1 week of study dose.
6. Non-smoking and no use of any tobacco or nicotine products (by declaration) for a period of at least 6 months prior to screening visit.
7. Be on no medication with potential to impair renal function (e.g., NSAIDs) or with ototoxic potential (e.g., quinine, salicylates, aminoglycosides).
8. Normal renal function (glomular filtration rate >60 mL/min) based on creatinine plasma concentration and the Modification of Diet in Renal Disease equation for estimated glomular filtration rate. Subjects with lower Modification of Diet in Renal Disease (MDRD) clearance can be included on the condition that they have a normal 24h creatinine clearance (determined by a 24h urine collection).
9. Negative human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) serology tests at screening.
10. No history of alcohol or drug of abuse (DOA). Negative urine test for DOA and alcohol breath test at screening and Day -1.
11. No personal history (or current) or hereditary hearing loss, persistent tinnitus, persistent vertigo, persistent imbalance, and persistent unsteadiness.
12. Body Mass Index (BMI) of 19.0 to 30.0 kg/m2 (inclusive); and a total body weight >50.0 kg (110 lbs) and <100.0 kg.

Subjects with any of the following characteristics/conditions will not be included in the study:

1. Subjects who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the Investigator, or subjects who are the Sponsor employees directly involved in the conduct of the study.
2. Concurrent participation or participation in another clinical trial within at least 5 tissue half-lives prior to dosing (calculated from the previous study's last dosing day). If the previous trial involved agents with delayed effects or prolonged metabolism, a 12 months interval is required.
3. Evidence or history of clinically relevant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies). This includes any acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational drug administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the subject inappropriate for entry into this study.
4. Presence of mitochondrial mutations making subject susceptible to aminoglycoside toxicity (A1555G, C1494T, T1095C, A827G, 1-BP DEL, 961T, C INS).
5. Subjects with any history of ear disease or surgeries, persistent dizziness or persistent tinnitus.
6. Subjects with any abnormality at screening, that indicates the presence of a vestibular pathology, conductive hearing loss or balance problem (by an ENT).

   Subjects with abnormalities in audiometry results at screening as follows: any pure tone threshold >55 dB and inter-ear difference in any frequency of >20 dB.

   Dizziness Handicap Inventory (DHI)-H score>16. Tinnitus Handicap Inventory (THI) H score >14.
7. History of regular alcohol consumption exceeding 14 drinks/week for females or 21 drinks/week for males (1 drink = 150 mL of wine or 360 mL of beer or 45 mL of hard liquor) within 6 months of screening.
8. Screening supine blood pressure (BP) ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at least 5 min of supine rest. If BP is ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), the BP should be repeated two more times and the average of the three BP values should be used to determine the subject's eligibility.
9. Screening supine 12-lead ECG demonstrating QTc >450 msec for men and >470 msec for women, or a QRS interval >120 msec. If QTc or QRS exceed these limits, the ECG should be repeated two more times and the average of the three QTc or QRS values should be used to determine the subject's eligibility.
10. Subjects with ANY abnormalities in clinical laboratory tests at screening, considered by the study physician as clinically relevant. In particular, subjects with alanine aminotransferase (ALT), aspartate aminotransferase (AST), serum creatinine and total bilirubin ≥1.5 upper limit of normal will be excluded.
11. Pregnant or breastfeeding female subjects.
12. Subjects who donated blood or received blood or plasma derivatives in the three months preceding study drug administration.
13. Unwilling or unable to comply with all scheduled visits, treatment plan, laboratory tests and other study procedures and the restrictions described in this protocol.
14. Known relevant allergy to any drug and/or aminoglycosides.
15. Subjects with an inability to communicate well with the Investigators and CPU staff (e.g., language problem, poor mental development).
16. Subjects with visual impairment or inability to read and comprehend the DHI and THI scales.
17. Subjects with any acute medical situation (e.g., acute infection) within 48 hours of study start, which is considered of significance by the Investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 0-10 days
  Incidence and characteristics of adverse events occurring following single doses of ELX-02
Pharmacokinetics: Maximum plasma concentration (Cmax) | 0-10 days
  Cmax will be determined for ELX-02 and an estimation of ELX-02 dose proportionality of PK parameters.
Pharmacokinetics: Time at which Cmax occurs (tmax) | 0-10 days
  tmax will be determined for ELX-02 and an estimation of ELX-02 dose proportionality of PK parameters.
Pharmacokinetics: Area under the plasma concentration-time curve calculated from time of administration to time 24h (AUC24h) | 0-10 days
  AUC24h will be determined for ELX-02 and an estimation of ELX-02 dose proportionality of PK parameters.
Pharmacokinetics: Area under the plasma concentration-time curve calculated from time of administration to time 48h (AUC48h) | 0-10 days
  AUC48h will be determined for ELX-02 and an estimation of ELX-02 dose proportionality of PK parameters.
Pharmacokinetics: Area under the concentration-time curve from time 0 extrapolated to infinity (AUCinf) | 0-10 days
  AUCinf will be determined for ELX-02 and an estimation of ELX-02 dose proportionality of PK parameters.
Pharmacokinetics: Mean residence time (MRT) | 0-10 days
  MRT will be determined for ELX-02 and an estimation of ELX-02 dose proportionality of PK parameters.
Pharmacokinetics: Elimination half-life (t1/2) | 0-10 days
  t1/2 will be determined for ELX-02 and an estimation of ELX-02 dose proportionality of PK parameters.
Pharmacokinetics: Volume of distribution (Vd/F) | 0-10 days
  Vd/F will be determined for ELX-02 and an estimation of ELX-02 dose proportionality of PK parameters.
Pharmacokinetics: Clearance (CL/F) | 0-10 days
  CL/F will be determined for ELX-02 and an estimation of ELX-02 dose proportionality of PK parameters.

CONTACTS AND LOCATIONS:
Locations (1):
- SGS Life Sciences, Clinical Pharmacology Unit, Antwerp, Belgium

REFERENCES:
- See also: Eloxx Pharmaceuticals Website — http://www.eloxxpharma.com